CLINICAL TRIAL: NCT03073863
Title: Statin Intensity, Achieved LDL Cholesterol, and Cardiovascular Outcome in Statin Therapy in Patients With Coronary Artery Disease (Post-hoc Study of TNT Trial)
Brief Title: Evaluation of Statin Mechanism Preventing Cardiovascular Disease by Post-hoc Analysis of Treating to New Targets Study
Acronym: TNTpost-hoc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Hong Seog Seo, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KUGH16082
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases
Keywords: LDL Cholesterol; Statin intensity; post hoc analysis; Achieved LDL Cholesterol level
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin 10mg (Active Comparator): 5006 patients received continuous medication with atorvastatin 10mg/day after run-in period.
  Interventions: Drug: Atorvastatin
- Atorvastatin 80mg (Experimental): 4995 patients received medication with atorvastatin 80mg/day after run-in period.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Analysis

SUMMARY:
Epidemiological studies have shown that serum cholesterol level is correlated with Cardiovascular Disease (CVD) risk, and that Cardiovascular Disease (CVD) risk increases with increasing LDL cholesterol levels. Fortunately, it has been confirmed that cholesterol-lowering therapy is effective in preventing Cardiovascular Disease (CVD), and cholesterol lowering with statin therapy is a primary strategy in the prevention of Cardiovascular Disease (CVD). Despite the fact that statins reduce both LDL cholesterol and future cardiovascular outcome, the association of statin intensity and the achieved level of LDL cholesterol with cardiovascular outcome has not been fully elucidated, because statins have pleiotropic effect as well as LDL lowering effect.

The effect of statin on future Cardiovascular (CV) outcome seems to be more associated with statin intensity relating pleiotropic effects rather than with achieved LDL cholesterol level, because LDL-lowering by inhibition of hepatic cholesterol synthesis is linked to reciprocal increment of cholesterol absorption from the intestine.

DETAILED DESCRIPTION:
It is easily extrapolated the relationship between LDL-C level and the incidence of Atherosclerotic Cardiovascular Disease (ASCVD) after statin therapy from the correlation between LDL-C level and the incidence of Atherosclerotic Cardiovascular Disease (ASCVD) in subjects without statin therapy and from the results of most lipid-lowering trials showing that 'the lower achieved LDL-C level, the better clinical outcomes. However, the association of statin intensity and the achieved level of LDL-C with cardiovascular outcome has not been fully elucidated, because the absolute amount of LDL cholesterol reduction is dependent not only on statin intensity, but also on inter-individual variation of statin responsiveness. In studies, the response to therapy with hypolipidemic agents shows considerable individual variation, and the use of the same dose of the same statin in different patients produces LDL-C decrease in a wide range from 8 to 55 %. These differences may be due to the interaction of environmental and genetic factors that affect drug bioavailability, receptor function or ligand structure and candidate gene analyses have found variants in known regulators of cholesterol metabolism such as HMGCR, Apolipoprotein E (APOE), PCSK9, Angiotensin Converting Enzyme (ACE), NPC1L1, and Low-Density Lipoprotein Receptor (LDLR) to be associated with statin response. Therefore, investigator suspects there could be some mistakes in interpreting the result of clinical trials with different intensities of statin. Actually, most of statin trials only compared the mean values of achieved LDL-C to the clinical outcomes in the statin therapy with different intensity, and there were few reports about the relationship between the individual values of achieved LDL-C and clinical outcomes in the statin therapy with same intensity. To accept the role of achieved LDL-C level for the prevention of Cardiovascular (CV) outcomes, it should still have a significant value after adjusting with statin intensity. In PROVE IT-Thrombolysis In Myocardial Infarction (TIMI) 22 study using either 80 mg of atorvastatin or 40 mg of pravastatin in Acute Coronary Syndrome (ACS) patients, IDEAL study with either 80 mg of atorvastatin or 20 mg of simvastatin in Acute Mycardial Infarction (AMI) patients, and TNT study with 80 mg of atorvastatin or 10 mg of atorvastatin in Coronary Artery Disease (CAD) patients, the authors demonstrated the relationships between the levels of achieved LDL-C after statin therapy and those between statin intensity and the risk of recurrent myocardial infarction or death from coronary causes separately. However, they did not report the relation between achieved LDL-C level and primary outcome after adjustment with statin intensity. Therefore, investigator think it may be inaccurate to determine the role of achieved LDL-C level in Atherosclerotic Cardiovascular Disease (ASCVD) prevention in clinical trials when those trials include the subjects with different intensity of statin therapy. Same phenomenon can also occur in meta-analysis of clinical trials with different statin intensity. Therefore, in Cholesterol Treatment Trialists' Collaboration (CTTC) meta-analyses, it should be reconsidered that the absolute amount of LDL-C reduction is dependent not only on statin intensity, but also on inter-individual variation of statin responsiveness.

All analyses will be performed on an intention-to-treat basis. Univariate analysis for each baseline characteristic of the patients, Cox proportional hazard model including age, sex, hypertension, diabetes, cardiovascular disease including coronary artery disease, cerebrovascular disease, peripheral artery disease, Congestive Heart Failure (CHF), achieved LDL cholesterol level, achieved C-Reactive Protein (CRP) level, statin intensity As in other studies using multiple doses of statin, investigator would like to evaluate the linear regression analysis between achieved LDL cholesterol level and CV outcome in total group, and it will show the correlation between them.

However, when investigator evaluates the linear regression analysis between achieved LDL cholesterol level and Cardiovascular (CV) outcome in the group treated with 10 mg of atorvastatin, it will show no relation between them, because of individual variability of LDL-C lowering effects by same statin.

The same result can be expected the relationship between achieved LDL cholesterol level and Cardiovascular (CV) outcome in the group treated with 80 mg of atorvastatin.

With the survival curve using Cox proportional hazard model for total Major Adverse Cardiac Events (MACE) and each component, investigator evaluates the impact of the followings:

1. Achieved LDL-C level ( quartiles)
2. Statin intensity
3. Achieved C-Reactive Protein (CRP) level ( quartiles)
4. Absolute mount of LDL-C lowering
5. Absolute mount of C-Reactive Protein (CRP) lowering
6. Other risk factors such as age, sex, hypertension, diabetes, hyperlipidemia, and etc.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 35 to 75 years of age
* Clinically evident Coronary Heart Disease (CHD), defined by one or more of the following:

  * previous myocardial infarction,
  * previous or current angina with objective evidence of CHD,
  * a history of coronary revascularization.

Exclusion Criteria:

* hypersensitivity to statins
* active liver disease or hepatic dysfunction defined as alanine aminotransferase or aspartate aminotransferase >1.5 times the upper limit of normal
* women who are pregnant or breastfeeding
* patients with nephrotic syndrome
* uncontrolled diabetes mellitus
* uncontrolled hypothyroidism
* uncontrolled hypertension at the screening visit;
* a Myocardial infarction (MI), coronary revascularization procedure or severe/unstable angina within 1 month of screening
* any planned surgical procedure for the treatment of atherosclerosis
* an ejection fraction <30%
* hemodynamically important valvular disease
* gastrointestinal disease limiting drug absorption or partial ileal bypass
* any nonskin malignancy, malignant melanoma or other survival-limiting disease
* unexplained creatine phosphokinase levels >6 times the upper limit of normal
* concurrent therapy with long-term immunosuppressants
* concurrent therapy with lipid-regulating drugs not specified as study treatment in the protocol
* history of alcohol abuse
* participation in another clinical trial concurrently or within 30 days before screening.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10001 (Actual)
Dates: Start 1998-04-03 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-01 (Actual)

PRIMARY OUTCOMES:
The Relation between achieved LDL cholesterol level and the occurence of a first major CV event after adjustment of statin intensity | Up to 6 years
  The effect of the achieved LDL cholesterol level on CV outcomes after adjustment of statin intensity.
  Definition of a first major cardiovascular event: death from CHD, nonfatal non-procedure-related myocardial infarction, resuscitation after cardiac arrest, or fatal or nonfatal stroke

SECONDARY OUTCOMES:
The Relation between statin intensity and the occurence of a first major CV event after adjustment of achieved LDL cholesterol level | Up to 6 years
  The effect of the statin intensity on CV outcomes after adjustment of achieved LDL cholesterol level
The Relation between th amount of LDL cholesterol level and the occurence of a first major CV event after adjustment of statin intensity | Up to 6 years
  The effect of LDL cholesterol lowering amount from baseline LDL-cholesterol on future CV outcome in statin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Seog Seo, MD, Principal Investigator — Korea University Guro Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaRosa JC, Grundy SM, Waters DD, Shear C, Barter P, Fruchart JC, Gotto AM, Greten H, Kastelein JJ, Shepherd J, Wenger NK; Treating to New Targets (TNT) Investigators. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med. 2005 Apr 7;352(14):1425-35. doi: 10.1056/NEJMoa050461. Epub 2005 Mar 8. PMID 15755765